CLINICAL TRIAL: NCT03978091
Title: A Phase 1, Open-Label Study in Healthy Adults to Evaluate the Safety and Pharmacokinetics of AVYCAZ(R) in Combination With Aztreonam (COMBINE)
Brief Title: A Trial to Evaluate the Pharmacokinetics and Safety of AVYCAZ(R) in Combination With Aztreonam
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0107; 5UM1AI104681-09 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2020-02-07

CONDITIONS: Bacterial Infection
Keywords: Aztreonam; Ceftazidime-Avibactam; Efficacy; Healthy; Pharmacokinetics; Population; Safety
MeSH Terms: conditions — Bacterial Infections | interventions — Aztreonam; avibactam, ceftazidime drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1 (Experimental): 2.5g dose of ceftazidime-avibactam (AVYCAZ) administered intravenously as a 2-hour infusion, every 8 hours for 7 days. N=8
  Interventions: Drug: Ceftazidime-Avibactam
- Arm 2 (Experimental): 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion once, then 0.32g dose per hour daily as a continuous infusion (7.5 g/day) for 7 days. N=8
  Interventions: Drug: Ceftazidime-Avibactam
- Arm 3 (Experimental): 2g dose of aztreonam (ATM) administered intravenously as a 2-hour infusion, every 6 hours for 7 days. N=8
  Interventions: Drug: AZACTAM
- Arm 4 (Experimental): 2g of ATM administered intravenously as a 2-hour infusion once, then 0.33g dose administered intravenously per hour, daily as a continuous infusion (8 g/day) for 7 days. N=8
  Interventions: Drug: AZACTAM
- Arm 5 (Experimental): 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion, every 8 hours for 7 days, and a 1.5g dose of ATM administered intravenously as a 2-hour infusion, every 6 hours for 7 days. N=8
  Interventions: Drug: AZACTAM; Drug: Ceftazidime-Avibactam
- Arm 6 (Experimental): 2.5 g dose of AVYCAZ administered intravenously as a 2-hour infusion every 8 hours for 7 days, and a 2g dose of ATM as a 2-hour infusion every 6 hours for 7 days. N=8
  Interventions: Drug: AZACTAM; Drug: Ceftazidime-Avibactam

INTERVENTIONS:
Drug: AZACTAM — A synthetic monobactam antibiotic originally isolated from Chromobacterium violaceum
  Arms: Arm 3; Arm 4; Arm 5; Arm 6
Drug: Ceftazidime-Avibactam — An antibacterial combination product containing ceftazidime and avibactam
  Arms: Arm 1; Arm 2; Arm 5; Arm 6

SUMMARY:
This is a Phase I, open-label, non-randomized, single center study in 48 healthy adult male and female subjects, aged 18 to 45 years. This study is aimed to investigate the safety and pharmacokinetics of ceftazidime-avibactam (AVYCAZ) combined with aztreonam (ATM), AVYCAZ alone, and ATM alone. The study will have 6 arms, arms 1-4 are the single drug administration treatment groups and will include AVYCAZ per label dosing, AVYCAZ as a continuous infusion (CI), ATM per label dosing, and ATM as a CI. Arms 5 and 6 are the two AVYCAZ and ATM combination drug administration treatment groups. The duration of subject participation will be up to 44 days, and the total length of the study will be 15 months. The primary objective of this study is to describe the safety of two dosing regimens of AVYCAZ combined with ATM relative to AVYCAZ alone, and ATM alone in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomized, single center study in 48 healthy adult male and female subjects, aged 18 to 45 years. This study is aimed to investigate the safety and pharmacokinetics of ceftazidime-avibactam (AVYCAZ) combined with aztreonam (ATM), AVYCAZ alone, and ATM alone. The study will have 6 arms, arms 1-4 are the single drug administration treatment groups and will include AVYCAZ per label dosing, AVYCAZ as a continuous infusion (CI), ATM per label dosing, and ATM as a continuous infusion (CI). Arms 5 and 6 are the two AVYCAZ and ATM combination drug administration treatment groups. The duration of subject participation will be up to 44 days, and the total length of the study will be 15 months. The primary objective of this study is to describe the safety of two dosing regimens of AVYCAZ combined with ATM relative to AVYCAZ alone, and ATM alone in healthy adult subjects. The secondary objectives of this study are to; 1) Characterize the PK profiles of two dosing regimens of AVYCAZ combined with ATM, AVYCAZ alone, and ATM alone at the population level in healthy adult subjects; 2) Characterize the PK profiles of two dosing regimens of AVYCAZ combined with ATM, AVYCAZ alone, and ATM alone following initiation of dosing on day 1 in healthy adult subjects; and 3) Characterize the PK profiles of two dosing regimens of AVYCAZ combined with ATM, AVYCAZ alone, and ATM alone following multiple daily dosing in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated written informed consent.
2. Be able to understand and willing to comply with study procedures, restrictions, and requirements, as determined by the Principal Investigator (PI).
3. Male and female volunteers aged 18 to 45 years inclusive.
4. Suitable veins for cannulation or repeated venipuncture.
5. Subject must be in good general health as judged by the investigator as determined by medical history, vital signs*, body mass index (BMI) and body weight**, clinical laboratory values***, and physical examination (PE).

   *Oral temp <38.0 degrees Celsius/100.4 degrees Fahrenheit; pulse 50 to 100 bpm; systolic blood pressure 90 to 140 mm Hg, and diastolic blood pressure 55 to 90 mmHg.

   **BMI between 19-33 kg/m^2 and body weight > / = 50 kg

   ***Clinical chemistry, hematology, coagulation and urinalysis results within the clinical laboratory reference ranges; clinical laboratory values outside these ranges, if considered by the site investigator to be clinically insignificant, are also acceptable
6. Sexually active female subjects must be of non-childbearing potential**** or must use a highly effective method of birth control*****.

   ****Non-childbearing potential is defined as being post-menopausal for at least 18 months or surgically sterile via hysterectomy, bilateral oophorectomy, or tubal sterilization.

   *****Sexually active female subjects of childbearing potential must avoid becoming pregnant by using one of the following acceptable methods of birth control for 30 days prior to study product dosing and must be maintained for 30 days after last dose of study product: Intrauterine contraceptive device; OR Approved hormonal contraceptives (such as birth control pills, skin patches, Implanon(R), Nexplanon(R), DepoProvera(R) or NuvaRing(R)); OR Birth control must be captured on the appropriate data collection form.
7. Sexually active male subjects must be vasectomized or agree to use barrier contraception (condom with spermicide) from first dose of study product until 30 days following the last dose of study product.
8. Nonsmokers defined as abstinence from cigarette smoking or use of nicotine-containing products for 6 months prior to enrollment into the study.

Exclusion Criteria:

1. History of any clinically significant (CS) disease or disorder, medical/surgical procedure, or trauma within 4 weeks prior to the first administration of study product(s)*.

   *In the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
2. History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Known history of a clinically important allergy/hypersensitivity to AVI, any monobactam, any beta-lactam and/or L-arginine.
4. Receipt of probenecid or furosemide within 14 days prior to study enrollment.
5. Receipt of any antibiotics within 14 days prior to study enrollment.
6. Receipt of prescription medications (except birth control pills or hormone replacement in females) within 14 days prior to study enrollment, unless in the opinion of site investigator the medication will not interfere with the study procedures or impact subject safety.
7. Receipt of non-antibiotic medications that interacts with OAT3** within 14 days prior to study enrollment.

   **Adefovir, Anagliptin, Baricitinib, Cefaclor, Cimetidine, Ciprofloxacin (Systemic), Clofarabine, Eluxadoline, Empagliflozin, Furosemide, Ketoprofen, Methotrexate, Mycophenolate, PEMEtrexed, Penicillin G (Parenteral/Aqueous), Penicillin G Benzathine, Penicillin G Procaine, Penicillin V Benzathine, Penicillin V Potassium, Zidovudine
8. Receipt of herbal and dietary supplements (including St. John's Wort) within 14 days prior to study enrollment.
9. ALT or AST laboratory value above the ULN as defined in the toxicity table.
10. Prolonged QTcF (> 450 msec) or shortened QTcF (< 340 msec) or family history of long QT syndrome. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG***.

    ***Abnormalities that may interfere with interpretation of QTc interval changes per the medical judgment of the PI.
11. Any positive result on screening for human immunodeficiency virus (HIV) serum hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) antibody.
12. Creatinine clearance equal or less than 80 mL/minute (measured by Cockcroft-Gault method).
13. History of Clostridium difficile infection in past 90 days.
14. Known or suspected history of drug or alcohol abuse within the last 5 years, as judged by the PI.
15. Positive screen for drugs of abuse, cotinine (nicotine), or alcohol at screening and at admission to the study site prior to the first administration of the study products(s).
16. Received a new chemical entity (compound not approved for marketing) or participated in a study that included drug treatment within 1 month of the first dose of study product(s) for study ****.

    ****Period of exclusion begins at the time of the last visit of the prior study.

    Note: subjects consented and screened, but not dosed in this study or a previous Phase I study will not be excluded.
17. Previous participation in the present study.
18. Involvement in the planning and/or conduct of the study.
19. Any ongoing/recent (during screening) medical complaints that may interfere with analysis of study data or are considered unlikely to comply with study procedures, restrictions, and requirements *****.

    *****Judgment by the PI that the subject should not participate in the study.
20. Known history of past or current epilepsy or seizure disorders, excluding febrile seizures of childhood.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult male and female subjects age 18-45, inclusively. Participants were enrolled between 09JUL2019 and 06NOV2020 and were recruited from the community around the clinical site.
Groups:
- AVYCAZ IV: 2.5g dose of ceftazidime-avibactam (AVYCAZ) administered intravenously as a 2-hour infusion, every 8 hours for 7 days.
  Ceftazidime-Avibactam: An antibacterial combination product containing ceftazidime and avibactam
- AVYCAZ CI: 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion once, then 0.32g dose per hour daily as a continuous infusion (CI) (7.5 g/day) for 7 days.
  Ceftazidime-Avibactam: An antibacterial combination product containing ceftazidime and avibactam
- ATM IV: 2g dose of aztreonam (ATM) administered intravenously as a 2-hour infusion, every 6 hours for 7 days.
  AZACTAM (aztreonam): A synthetic monobactam antibiotic originally isolated from Chromobacterium violaceum
- ATM CI: 2g of ATM administered intravenously as a 2-hour infusion once, then 0.33g dose administered intravenously per hour, daily as a continuous infusion (CI) (8 g/day) for 7 days.
  AZACTAM: A synthetic monobactam antibiotic originally isolated from Chromobacterium violaceum
- AVYCAZ + ATM 1.5: 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion, every 8 hours for 7 days, and a 1.5g dose of ATM administered intravenously as a 2-hour infusion, every 6 hours for 7 days.
  AZACTAM: A synthetic monobactam antibiotic originally isolated from Chromobacterium violaceum
  Ceftazidime-Avibactam: An antibacterial combination product containing ceftazidime and avibactam
- AVYCAZ + ATM 2.0: 2.5 g dose of AVYCAZ administered intravenously as a 2-hour infusion every 8 hours for 7 days, and a 2g dose of ATM as a 2-hour infusion every 6 hours for 7 days.
  AZACTAM: A synthetic monobactam antibiotic originally isolated from Chromobacterium violaceum
  Ceftazidime-Avibactam: An antibacterial combination product containing ceftazidime and avibactam
Period: Overall Study
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 7 | 7 | 8
Not Completed | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes the number of participants in the safety population.
Groups:
- AVYCAZ IV: 2.5g dose of ceftazidime-avibactam (AVYCAZ) administered intravenously as a 2-hour infusion, every 8 hours for 7 days.
- AVYCAZ CI: 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion once, then 0.32g dose per hour daily as a continuous infusion (CI) (7.5 g/day) for 7 days.
- ATM IV: 2g dose of aztreonam (ATM) administered intravenously as a 2-hour infusion, every 6 hours for 7 days.
- ATM CI: 2g of ATM administered intravenously as a 2-hour infusion once, then 0.33g dose administered intravenously per hour, daily as a continuous infusion (CI) (8 g/day) for 7 days.
- AVYCAZ + ATM 1.5: 2.5g dose of AVYCAZ administered intravenously as a 2-hour infusion, every 8 hours for 7 days, and a 1.5g dose of ATM administered intravenously as a 2-hour infusion, every 6 hours for 7 days.
- AVYCAZ + ATM 2.0: 2.5 g dose of AVYCAZ administered intravenously as a 2-hour infusion every 8 hours for 7 days, and a 2g dose of ATM as a 2-hour infusion every 6 hours for 7 days.
- Total: Total of all reporting groups
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 8 | 8 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (5.5) | 36.4 (7.0) | 34.5 (5.9) | 30.8 (6.5) | 28.5 (3.8) | 33.8 (4.6) | 33.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 5 | 4 | 4 | 24
  Male | 4 | 6 | 3 | 3 | 4 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 1 | 1 | 2 | 8
  Not Hispanic or Latino | 8 | 7 | 5 | 7 | 7 | 6 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 3 | 7 | 4 | 4 | 29
  White | 2 | 2 | 2 | 1 | 1 | 2 | 10
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 48
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.74 (2.92) | 27.65 (3.44) | 26.16 (3.52) | 25.38 (4.09) | 25.55 (3.33) | 28.31 (4.58) | 26.46 (3.66)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Grade 2 (Moderate) or Higher Treatment-emergent Adverse Event
Description: Adverse events include local and systemic reactions. All Grade 2 (moderate) adverse events were reported, regardless of relationship to study product. Number of participants with an AE are summarized by MedDRA system organ class (SOC). Each participant is only counted once per SOC.
Time Frame: Day 1 through Day 11
Population: The safety population includes all participants who received any amount of study product (started first infusion).
Measure: Count of Participants; unit: Participants
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants
  Cardiac Disorders | 1 | 0 | 0 | 1 | 1 | 0
  Eye disorders | 0 | 0 | 0 | 1 | 0 | 0
  General disorders and administration site conditions | 0 | 0 | 1 | 0 | 0 | 0
  Infections and infestations | 0 | 0 | 1 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 0 | 0 | 0 | 1
  Investigations | 3 | 1 | 3 | 5 | 4 | 4
  Nervous system disorders | 0 | 0 | 1 | 1 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Accumulation Ratio for AUC (Area Under the Plasma Concentration-time Curve of Study Drug) [RAUC]
Description: Mean and standard deviation (SD) of the RAUC PK parameter were estimated for ceftazidime, avibactam, and/or aztreonam by dividing the AUC(0-8) (avibactam and ceftazidime) or AUC(0-6) (aztreonam) on Day 7 by the AUC(0-Tau) on Day 1. AUC(0-8) and AUC(0-6) (µg*hr/mL) on Day 7 and AUC(0-Tau) (µg*hr/mL) on Day 1 were estimated from plasma concentration-time data using Non-compartmental analysis with the linear trapezoidal linear interpolation method for AVYCAZ IV, ATM IV, AVYCAZ + ATM 1.5, and AVYCAZ + ATM 2.0.
Time Frame: Day 1 and Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The AVYCAZ + ATM 1.5 arm consists of 4 participants as 4 participants missed aztreonam doses on day 7. The AVYCAZ CI and ATM CI arms consist of 0 participants as AUC(0-Tau) was not collected on Day 1 due to the study drug being administered as a continuous infusion.
Measure: Mean (Standard Deviation); unit: Accumulation ratio
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 0 | 8 | 0 | 4 | 8
Accumulation ratio
  Avibactam: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 8
  Avibactam | 0.87 (0.12) |  |  |  | 0.80 (0.03) | 0.82 (0.06)
  Ceftazidime: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 8
  Ceftazidime | 0.98 (0.12) |  |  |  | 0.95 (0.04) | 0.95 (0.05)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 0.90 (0.07) |  | 0.91 (0.04) | 0.94 (0.05)

3. Secondary Outcome: Accumulation Ratio for Cmax (Maximum Plasma Concentration) (RCmax)
Description: Mean and standard deviation (SD) of the RCmax PK parameter were estimated for ceftazidime, avibactam, and/or aztreonam by dividing the Cmax on Day 7 by the Cmax on Day 1. Cmax (ug/mL) was estimated from plasma concentration-time data using Non-compartmental analysis for AVYCAZ IV, ATM IV, AVYCAZ + ATM 1.5, and AVYCAZ + ATM 2.0.
Time Frame: Day 1 and Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The AVYCAZ + ATM 1.5 arm consists of 4 participants as 4 participants missed aztreonam doses on day 7. The AVYCAZ CI and ATM CI arms consist of 0 participants as this data was not collected in arms where the study drug was administered as a continuous infusion.
Measure: Mean (Standard Deviation); unit: Accumulation ratio
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 0 | 8 | 0 | 4 | 8
Accumulation ratio
  Avibactam: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 8
  Avibactam | 0.88 (0.18) |  |  |  | 0.83 (0.05) | 0.91 (0.08)
  Ceftazidime: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 8
  Ceftazidime | 0.96 (0.20) |  |  |  | 0.96 (0.06) | 1.01 (0.11)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 0.88 (0.07) |  | 0.95 (0.05) | 0.97 (0.11)

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve of Study Drug From Time of Dosing Extrapolated to Infinity [AUC(0-Inf)]
Description: Mean and standard deviation (SD) of the AUC(0-inf) (µg*hr/mL) PK parameter were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. Participants in the ATM CI arm do not have data because dosing for all participants was stopped prior to Day 7, so their PK data was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 8
µg*hr/mL
  Avibactam: number analyzed (Participants) | 8 | 7 | 0 | 0 | 4 | 8
  Avibactam | 32.10 (3.73) | 42.40 (7.17) |  |  | 39.10 (4.57) | 36.10 (6.17)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Ceftazidime | 235.00 (25.80) | 308.00 (63.30) |  |  | 277.00 (27.50) | 249.00 (26.40)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 263.00 (38.80) |  | 245.00 (23.50) | 317.00 (47.70)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve Data of Study Drug During the Dosing Interval on Day 1 [AUC(0-Tau)]
Description: Mean and standard deviation (SD) of the AUC(0-Tau) (µg*hr/mL) PK parameter were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis using linear trapezoidal linear interpolation method for AVYCAZ IV, ATM IV, AVYCAZ + ATM 1.5, and AVYCAZ + ATM 2.0. AVYCAZ CI and ATM CI were not reported.
Time Frame: Day 1
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The AVYCAZ CI and ATM CI arms consist of 0 participants as AUC(0-Tau) was not collected on Day 1 due to the study drug being administered as a continuous infusion.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 8
µg*hr/mL
  Avibactam: number analyzed (Participants) | 8 | 0 | 0 | 0 | 8 | 8
  Avibactam | 35.80 (5.96) |  |  |  | 44.00 (7.10) | 42.40 (7.16)
  Ceftazidime: number analyzed (Participants) | 8 | 0 | 0 | 0 | 8 | 8
  Ceftazidime | 223.00 (33.90) |  |  |  | 255.00 (34.30) | 241.00 (33.10)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 8 | 8
  Aztreonam |  |  | 266.00 (36.10) |  | 221.00 (32.70) | 295.00 (41.30)

6. Secondary Outcome: Incidence of Treatment-emergent Adverse Events, by System Organ Class (SOC) and Maximum Severity Level
Description: Number of participants with an AE are summarized by MedDRA system organ class (SOC) and severity. Each participant is only counted once at the highest severity recorded. For clinical laboratory tests, mild abnormal laboratory values that were not, in the investigator's opinion, medically significant were not reported as adverse events.
Time Frame: Day 1 through Day 14
Population: The safety population includes all participants who received any amount of study product (started first infusion).
Measure: Count of Participants; unit: Participants
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants
  Cardiac Disorders: Mild | 2 | 2 | 4 | 1 | 3 | 2
  Cardiac Disorders: Moderate | 1 | 0 | 0 | 0 | 1 | 0
  Cardiac Disorders: Severe | 0 | 0 | 0 | 1 | 0 | 0
  Cardiac Disorders: None | 5 | 6 | 4 | 6 | 4 | 6
  Eye disorders: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: Moderate | 0 | 0 | 0 | 1 | 0 | 0
  Eye disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: None | 8 | 8 | 8 | 7 | 8 | 8
  Gastrointestinal Disorders: Mild | 3 | 1 | 2 | 0 | 5 | 3
  Gastrointestinal Disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal Disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal Disorders: None | 5 | 7 | 6 | 8 | 3 | 5
  General disorders and administration site conditions: Mild | 2 | 2 | 3 | 2 | 3 | 4
  General disorders and administration site conditions: Moderate | 0 | 0 | 1 | 0 | 0 | 0
  General disorders and administration site conditions: Severe | 0 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditions: None | 6 | 6 | 4 | 6 | 5 | 4
  Infections and infestations: Mild | 0 | 0 | 0 | 0 | 1 | 0
  Infections and infestations: Moderate | 0 | 0 | 1 | 0 | 0 | 0
  Infections and infestations: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations: None | 8 | 8 | 7 | 8 | 7 | 8
  Injury, poisoning and procedural complications: Mild | 0 | 0 | 2 | 0 | 1 | 0
  Injury, poisoning and procedural complications: Moderate | 0 | 0 | 0 | 0 | 0 | 1
  Injury, poisoning and procedural complications: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications: None | 8 | 8 | 6 | 8 | 7 | 7
  Investigations: Mild | 1 | 4 | 3 | 2 | 4 | 4
  Investigations: Moderate | 2 | 1 | 2 | 3 | 3 | 4
  Investigations: Severe | 1 | 0 | 1 | 2 | 1 | 0
  Investigations: None | 4 | 3 | 2 | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders: Mild | 1 | 1 | 1 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: None | 7 | 7 | 7 | 8 | 8 | 8
  Nervous system disorders: Mild | 1 | 1 | 1 | 0 | 2 | 0
  Nervous system disorders: Moderate | 0 | 0 | 1 | 1 | 0 | 0
  Nervous system disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders: None | 7 | 7 | 6 | 7 | 6 | 8
  Renal and urinary disorders: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Renal and urinary disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Renal and urinary disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Renal and urinary disorders: None | 8 | 8 | 8 | 8 | 8 | 7
  Respiratory, thoracic and mediastinal disorders: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: Moderate | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: None | 8 | 8 | 8 | 8 | 7 | 8
  Skin and subcutaneous tissue disorders: Mild | 1 | 1 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: None | 7 | 7 | 8 | 8 | 8 | 8
  Vascular disorders: Mild | 1 | 1 | 3 | 0 | 1 | 2
  Vascular disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: None | 7 | 7 | 5 | 8 | 7 | 6

7. Secondary Outcome: Maximum Plasma Concentration of Study Drug After the First Dose (Cmax)
Description: Mean and standard deviation (SD) of the Cmax (ug/mL) PK parameter after the first dose were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 1
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
ug/mL
  Avibactam: number analyzed (Participants) | 8 | 8 | 0 | 0 | 8 | 8
  Avibactam | 12.40 (2.38) | 13.10 (2.20) |  |  | 15.80 (3.04) | 14.30 (2.69)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 8 | 8
  Ceftazidime | 67.90 (14.00) | 71.20 (11.80) |  |  | 82.70 (18.50) | 70.30 (12.70)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 8 | 8 | 8
  Aztreonam |  |  | 89.10 (10.40) | 93.80 (4.98) | 71.20 (12.80) | 93.20 (15.80)

8. Secondary Outcome: Maximum Plasma Concentration of Study Drug Following Multiple Daily Dosing (Cmax)
Description: Mean and standard deviation (SD) of the Cmax (ug/mL) PK parameter following multiple daily dosing were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 8
ug/mL
  Avibactam: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Avibactam | 10.70 (2.52) | 4.58 (0.74) |  |  | 14.20 (1.75) | 12.80 (2.03)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Ceftazidime | 63.60 (12.60) | 31.80 (6.31) |  |  | 88.20 (12.40) | 69.80 (8.31)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 78.40 (9.38) |  | 74.40 (9.14) | 90.30 (16.70)

9. Secondary Outcome: Minimum Plasma Concentration of Study Drug at the End of the Dosing Interval on Day 7 (Cmin)
Description: Mean and standard deviation (SD) of the Cmin (ug/mL) PK parameter were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis for AVYCAZ IV, ATM IV, AVYCAZ + ATM 1.5, and AVYCAZ + ATM 2.0. Cmin was not provided on day 7 because it was the last dosage of the study product administered; Cmin was therefore not calculated for this terminal elimination profile since the minimum concentration after a final dose would only reflect the last time point after Cmax that a blood sample is obtained, or the assay's limit of quantitation. It is therefore not comparable to Cmin calculated on prior days.
Time Frame: Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. Zero participants have data because this analysis was not performed.
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Minimum Plasma Concentration of Study Drug Following Multiple Daily Dosing on Day 1 (Cmin)
Description: Mean and standard deviation (SD) of the Cmin (ug/mL) PK parameter were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis for AVYCAZ IV, ATM IV, AVYCAZ + ATM 1.5, and AVYCAZ + ATM 2.0.
Time Frame: Day 1
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The AVYCAZ CI and ATM CI arms consist of 0 participants as this data was not collected in arms where the study drug was administered as a continuous infusion.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 8
ug/mL
  Avibactam: number analyzed (Participants) | 8 | 0 | 0 | 0 | 8 | 8
  Avibactam | 0.52 (0.20) |  |  |  | 0.74 (0.40) | 0.72 (0.29)
  Ceftazidime: number analyzed (Participants) | 8 | 0 | 0 | 0 | 8 | 8
  Ceftazidime | 5.52 (1.20) |  |  |  | 6.29 (2.58) | 6.28 (1.54)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 8 | 8
  Aztreonam |  |  | 13.90 (2.84) |  | 13.30 (1.91) | 18.90 (3.99)

11. Secondary Outcome: Renal Clearance of Study Drug (CLR)
Description: Mean and standard deviation (SD) of the CLR (L/h) PK parameter were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma and urine concentration-time data using Non-compartmental analysis. Renal clearance was calculated as Ae(0-8)/AUC(0-8) for ceftazidime and avibactam and as AE(0-4)/AUC(0-4) for aztreonam where Ae(0-8) and Ae(0-4) are the amounts of study drug excreted into the urine from time of dosing to 8 or 4 h post-dose, respectively, and AUC(0-8) and AUC(0-4) are the areas under the plasma concentration-time curve from time of dosing to 8 or 4 h post-dose, respectively.
Time Frame: Day 1
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The AVYCAZ CI and AVYCAZ + ATM 2.0 arms consist of 7 participants due to participants missing the urine collection interval.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
L/h
  Avibactam: number analyzed (Participants) | 8 | 7 | 0 | 0 | 8 | 7
  Avibactam | 11.10 (2.58) | 11.70 (2.61) |  |  | 11.40 (2.36) | 14.70 (5.35)
  Ceftazidime: number analyzed (Participants) | 8 | 7 | 0 | 0 | 8 | 7
  Ceftazidime | 5.70 (1.23) | 6.92 (1.71) |  |  | 7.10 (1.09) | 9.42 (3.00)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 8 | 8 | 7
  Aztreonam |  |  | 4.25 (0.91) | 3.90 (0.97) | 4.61 (1.66) | 4.50 (1.08)

12. Secondary Outcome: Concentration of Study Drug at Steady State After Continuous Infusion (Css)
Description: Mean and standard deviation (SD) of the Css (ug/mL) PK parameter were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data for AVYCAZ CI and ATM CI.
Time Frame: Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 0 | 8 | 0 | 8 | 0 | 0
ug/mL
  Avibactam: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0
  Avibactam |  | 4.34 (1.80) |  |  |  |
  Ceftazidime: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0
  Ceftazidime |  | 27.60 (11.40) |  |  |  |
  Aztreonam: number analyzed (Participants) | 0 | 0 | 0 | 8 | 0 | 0
  Aztreonam |  |  |  | 58.80 (6.05) |  |

13. Secondary Outcome: Total Body Plasma Clearance of Study Drug (CL)
Description: Mean and standard deviation (SD) of the CL (L/h) PK parameter were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. The ATM CI arm consists of 0 participants as dosing for all was stopped prior to Day 7. The AVYCAZ + ATM 1.5 arm consists of 4 participants as they missed doses on day 7. One participant in AVYCAZ CI for avibactam had an elimination parameter that did not meet acceptance criteria and was excluded.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 8
L/h
  Avibactam: number analyzed (Participants) | 8 | 7 | 0 | 0 | 4 | 8
  Avibactam | 15.80 (1.85) | 12.20 (2.38) |  |  | 12.90 (1.59) | 14.30 (2.85)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Ceftazidime | 8.59 (0.95) | 6.80 (1.59) |  |  | 7.26 (0.68) | 8.13 (1.01)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 7.74 (1.07) |  | 6.18 (0.57) | 6.47 (1.20)

14. Secondary Outcome: Time of Cmax (Maximum Plasma Concentration) of Study Drug After the First Dose (Tmax)
Description: Mean and standard deviation (SD) of the Tmax (h) PK parameter after the first dose were estimated from the Day 1 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
h
  Avibactam: number analyzed (Participants) | 8 | 8 | 0 | 0 | 8 | 8
  Avibactam | 1.89 (0.35) | 2.00 (0.00) |  |  | 1.81 (0.27) | 1.99 (0.01)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 8 | 8
  Ceftazidime | 2.06 (0.42) | 2.06 (0.18) |  |  | 1.93 (0.33) | 1.93 (0.18)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 8 | 8 | 8
  Aztreonam |  |  | 1.94 (0.18) | 2.00 (0.01) | 1.99 (0.02) | 2.06 (0.18)

15. Secondary Outcome: Time to Cmax (Maximum Plasma Concentration) of Study Drug Following Multiple Daily Dosing (Tmax)
Description: Mean and standard deviation (SD) of the Tmax (h) PK parameter following multiple daily dosing were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 7
Population: The PK population includes all participants who received at least one dose of study drug and had at least one quantifiable plasma or urine concentration of ceftazidime, avibactam, or aztreonam. Participants in the ATM CI arm do not have data because dosing for all participants was stopped prior to Day 7, so their PK data was excluded from the analysis. The AVYCAZ + ATM 1.5 arm consists of 4 participants as 4 participants missed aztreonam doses on day 7.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 8
h
  Avibactam: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Avibactam | 1.82 (0.27) | 2.85 (2.59) |  |  | 1.99 (0.02) | 1.88 (0.23)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Ceftazidime | 2.14 (0.35) | 2.25 (2.06) |  |  | 1.86 (0.25) | 1.88 (0.23)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 2.00 (0.00) |  | 1.99 (0.02) | 2.00 (0.04)

16. Secondary Outcome: Volume of Distribution of Study Drug at Steady-state Based on the Last Observed Concentration (Vss)
Description: Mean and standard deviation (SD) of the Vss (L) PK parameter were estimated from the Day 7 ceftazidime, avibactam, and/or aztreonam plasma concentration-time data using Non-compartmental analysis.
Time Frame: Day 7
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
Number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 8
L
  Avibactam: number analyzed (Participants) | 8 | 7 | 0 | 0 | 4 | 8
  Avibactam | 25.90 (5.26) | 17.40 (4.91) |  |  | 18.50 (4.48) | 24.30 (6.65)
  Ceftazidime: number analyzed (Participants) | 8 | 8 | 0 | 0 | 4 | 8
  Ceftazidime | 19.90 (3.86) | 12.60 (3.17) |  |  | 14.50 (2.86) | 19.20 (4.27)
  Aztreonam: number analyzed (Participants) | 0 | 0 | 8 | 0 | 4 | 8
  Aztreonam |  |  | 14.30 (1.86) |  | 11.50 (2.14) | 13.80 (3.17)

ADVERSE EVENTS:
Time Frame: Local and systemic adverse events (AEs) and serious adverse events (SAEs) were recorded occurring from first dose of study product day 1 through the final visit, up to 14 days following the first dose.
Arm/Group | AVYCAZ IV | AVYCAZ CI | ATM IV | ATM CI | AVYCAZ + ATM 1.5 | AVYCAZ + ATM 2.0
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 6/8 | 7/8 | 8/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVYCAZ IV (N=8) | AVYCAZ CI (N=8) | ATM IV (N=8) | ATM CI (N=8) | AVYCAZ + ATM 1.5 (N=8) | AVYCAZ + ATM 2.0 (N=8)
Bradycardia (Cardiac disorders) | 2 (4) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Infusion site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Infusion site phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal bruit (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 3 (3) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 4 (4) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03978091/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03978091/SAP_002.pdf
  • Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03978091/ICF_000.pdf